CLINICAL TRIAL: NCT06160219
Title: Prophylactic Use of Hydroxycobolamin in the Prevention of Vasoplegic Syndrome in Adult Patients Undergoing Cardiopulmonary Bypass
Brief Title: Prophylactic Use of Hydroxycobolamin in Vasoplegic Syndrome in Adult Patients Undergoing Cardiopulmonary Bypass
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Salah Eldin Mahmoud Badre, Associate Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU R46/2019
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Vasoplegic Syndrome
MeSH Terms: conditions — Vasoplegia | interventions — Hydroxocobalamin; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: At the end of CPB, the patients will be assigned randomly into 2 groups by using computer generated random numbers sequences and sealed envelopes.
  Group (OH CO): 30 patients will receive hydroxycobolamin (Cyanokit) 5 gm intravenously(iv) through the central venous catheter as bolus over 15 min reconstituted in 200 ml of NS.
  Group (C) control: 30 patients will receive 200ml of NS over 15 min iv.
  Primary outcome will be change in MAP between baseline and all time points (30 & 60 min after CPB initiation) and (30 & 60 min after CPB separation) between the two groups and within the same group.
  Secondary outcomes were:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (OH CO) (Active Comparator): Group (OH CO): 30 patients will receive hydroxycobolamin (Cyanokit) 5 gm intravenously(iv) through the central venous catheter as bolus over 15 min reconstituted in 200 ml of NS.
  Interventions: Drug: Hydroxycobalamin
- Group (C) control (Placebo Comparator): Group (C) control: 30 patients will receive 200ml of NS over 15 min iv.
  Interventions: Drug: Hydroxycobalamin

INTERVENTIONS:
Drug: Hydroxycobalamin — prophylactic use of hydroxycobalamin in vasoplegia in high risk patients undergoing cardiac surgeries
  Other Names: Synthetic vitamin B12 ( cyanokit)

SUMMARY:
Several studies have described the use of alternative drugs as methylene blue (MB) (3) other than the standard limited options of the use of vasopressors and systemic corticosteroids (4) especially in the face of increasing incidence of vasoplegic syndrome. Hydroxycobolamin (HCO) has been used for treating cyanide poisoning for more than 40 years. Persistant and significant hypertension occurred as a result of the ability of (HCO) to bind nitric oxide (NO) to form nitrocobalamin.

In this prospective randomized controlled trial, we hypothesized that the prophylactic use of HCO in high risk patients after CPB may decrease the incidence of vasoplegia.

DETAILED DESCRIPTION:
Patients and methods

This randomized placebo-controlled single -center study will be conducted in Ain Shams University Hospital from May 2019 till October 2022. Patients undergoing Cardiopulmonary bypass grafting (CABG) and/or valve surgery will be approached by their anesthesia providers. Those who will be accepted to participate in the study were screened for inclusion and exclusion criteria on the day of the surgery or one day before. Informed consent will be taken from all participants by anesthesia providers. The duration of the study will be from the start of cardiac surgical procedure till after separation from CPB by 60 minutes.

Patients will be included in the study are aged from18- 60 yrs old undergoing CABG and/or valve surgery on CPB and have 2 or more preoperative risk factors for Vasoplegia including

* Using preoperative beta blocker (BB) or Angiotensin converting enzyme inhibitor (ACEI).
* preoperative EF < 35%
* History of thyroid disease
* Preoperative diuretics

Exclusion criteria are:

1. Emergency surgery
2. Severe renal Insufficiency (preoperative Cr > 1.8 mg / dL)
3. Severe hepatic disease (preoperative diagnosis of liver cirrhosis or recent elevated liver function tests
4. Pregnant or woman of child bearing potential
5. Know hypersensitivity to hydroxycobolamin

Preoperative data will be obtained from the medical records and verified with the patients; sex, age, Body surface index (BSI) , height and weight, type of surgery , preoperative use of ;ACEI- BB- calcium channel blocker (CCB) - amiodarone, mean arterial blood pressure (MAP), preoperative Ejection fraction (EF). Anesthesia will be induced in all patients and maintained by using midazolam, fentanyl, propofol, sevoflurane, pancurium.

* All patients were monitored with the routine monitoring of all cardiac patients which included: MAP in mmHg, oxygen saturation (SaO2), central venous pressure (CVP) in cmH2o, electrocardiography (ECG), Cardiac output (CO) L/min, arterial blood gases (ABG) measuring; PH, PaCo2, HCO3, lactate during the pre- during- post CPB, trans-esophageal echocardiography (TEE) measuring CO, CI, LVEF, SVR ( dyne.s/cm5)=MAP-CVP/CO✖ 800, SVRI= MAP-CVP/ CI ✖ 800.

Vasopressors in the form of norepinephrine will be started and titrated to maintain MAP >60 mmHg in the pre- during - post CPB period.

The total doses of norepinephrine and epinephrine (if needed) in (µg/kg/min) will be recorded on the anesthesia record by anesthesia providers. After induction of CPB all patients undergo non pulsatile hypothermia (32-34 0C) CPB with a membrane oxygenator and the arterial line filter. Priming of CPB will be done by crystalloids and serial HCT level were at >18%. The flow rate on CPB was 2- 2.5L/ min/ m2 to maintain the MAP 50-80 mmHg. Blood gases samples will be measured every 30 min to maintain arterial CO2 of 35-40 mmHg uncorrected for temperature (alpha stat) and the partial pressure of O2 (150-250 mmHg). Hemodynamics will be recorded every 30 min intervals and stored into the anesthesia record. The time of CPB and cross clamping time will be recorded.

At the end of CPB, the patients will be assigned randomly into 2 groups by using computer generated random numbers sequences and sealed envelopes.

Group (OH CO): 30 patients will receive hydroxycobolamin (Cyanokit) 5 gm intravenously(iv) through the central venous catheter as bolus over 15 min reconstituted in 200 ml of NS.

Group (C) control: 30 patients will receive 200ml of NS over 15 min iv.

Primary outcome will be change in MAP between baseline and all time points (30 & 60 min after CPB initiation) and (30 & 60 min after CPB separation) between the two groups and within the same group.

Secondary outcomes were:

1. Change in SVR between baseline and all time points (30 & 60 min after CPB initiation) and (30 & 60 min after CPB separation) between the 2 groups and within the same group.
2. Number of patients who needed norepinephrine ≥ 0.5µg/kg/min ± epinephrine as inotropic support during weaning from CPB.
3. Incidence of vasoplegic syndrome occurrence which is defined as occurrence of one or more of these parameters: systemic vascular resistance of ≤ 800 dyne/ s/ cm, an MAP of ≤ 60 to 65 mm Hg, a cardiac index of ≥ 2.5 to 3 L/ min/ m2, a requirement for at least one or more high-dose of vasopressors (ie, norepinephrine >0.05 μg / kg/ min).
4. Number of patients who developed norepinephrine refractory vasoplegia ( needed epinephrine as another inotropic support)
5. Number of patients developed multiorgan failure in ICU
6. Mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study are aged from18- 60 yrs old undergoing CABG and/or valve surgery on CPB and have 2 or more preoperative risk factors for Vasoplegia,
* Using preoperative beta blocker (BB) or Angiotensin converting enzyme inhibitor (ACEI).
* preoperative EF < 35%
* History of thyroid disease
* Preoperative diuretics

Exclusion Criteria:

* Exclusion criteria are:

  1. Emergency surgery
  2. Severe renal Insufficiency (preoperative Cr > 1.8 mg / dL)
  3. Severe hepatic disease (preoperative diagnosis of liver cirrhosis or recent elevated liver function tests
  4. Pregnant or woman of child bearing potential
  5. Know hypersensitivity to hydroxycobolamin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
change in systemic vascular resistance | within 30 and 60 minutes
  Primary outcome will be change in MAP between baseline and all time points (30 & 60 min after CPB initiation) and (30 & 60 min after CPB separation) between the two groups and within the same group.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Badre, MD, Principal Investigator — Associate Professor of Anesthesia and ICU , Ain Shams University
Locations (1):
- AinShams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: within 6 months for 4 years time
Access Criteria: all IPD data of protocol, results and discussion.